CLINICAL TRIAL: NCT06075043
Title: A Multicenter, Randomized, Open-label Study of AND017 for the Treatment of Anemia of Cancer in Patients Not Receiving Chemotherapy
Brief Title: A Study of AND017 to Treat Cancer Related Anemia in Patients Not Receiving Chemotherapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kind Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AND017-CRA-202
Record Dates: First submitted 2023-03-22; First posted 2023-10-10 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Cancer-Related Anemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AND017 Dose A three times weekly (Experimental)
  Interventions: Drug: AND017
- AND017 Dose B three times weekly (Experimental)
  Interventions: Drug: AND017
- AND017 Dose C three times weekly (Experimental)
  Interventions: Drug: AND017

INTERVENTIONS:
Drug: AND017 — Oral administration of AND017 capsules three times per week

SUMMARY:
The purpose of this study is to determine the safety and efficacy of various doses of AND017 after 6 weeks of treatment in subjects with anemia of cancer who are not receiving chemotherapy.

ELIGIBILITY:
Main Inclusion Criteria:

1. Non-myeloid malignancy diagnosed by cytology/histology.
2. ECOG score 0-2 and expected survival of 6 months or more.
3. The mean value of hemoglobin at screening test and one follow-up test (more than one week between tests) was <10.0 g/dL, with a difference of ≤1.0 g/dL between the two tests.
4. Adequate hepatic and renal function.

   * Total bilirubin < 1.5 x upper limit of normal (ULN).
   * Subjects with Gilbert's syndrome (unconjugated hyperbilirubinemia) have a total bilirubin < 3 x ULN.
   * Aspartate aminotransferase (AST)
   * Alanine aminotransferase (ALT) <2.5 x ULN
   * eGFR >60 mL/min/1.73

Exclusion Criteria:

1. Received chemotherapy, radiotherapy, and other, e.g., immunosuppressive, targeted drug therapy that has a suppressive effect on the bone marrow within 1 month prior to randomization or planned during the trial.
2. A medical history of significant liver disease or active liver disease.
3. A previous history of pure red blood cell remittance
4. A combination of hereditary anemia, iron-granulocytic anemia, acute blood loss, active bleeding (three consecutive positive fecal occult bloods or clinical judgment of the investigator), hemolysis and other conditions that can cause anemia such as iron, folic acid or vitamin B12 deficiency
5. Active infection or inflammatory disease requiring systemic anti-infective therapy within 1 week prior to the first dose, including concurrent autoimmune diseases with inflammatory symptoms (e.g., generalized erythema, ankylosing spondylitis, rheumatoid arthritis, psoriatic arthritis, dry syndrome, celiac disease, etc.)
6. Concurrent retinal neovascularization requiring treatment (diabetic proliferative retinopathy, age-related exudative macular degeneration, retinal vein occlusion, macular edema, etc.).
7. clinically significant bleeding (including the need for blood transfusion or a drop in hemoglobin ≥ 2 g/dL) within 4 weeks prior to the first dose, or a bleeding constitutional or bleeding risk that has not been medically or surgically corrected
8. uncontrolled hypertension (more than one-third of identifiable diastolic blood pressure values > 90 mmHg and/or systolic blood pressure ≥ 160 mmHg at 16 weeks prior to and including screening testing)
9. concurrent congestive heart failure (New York Heart Association [NYHA] class III or higher)
10. clinically significant ECG abnormalities at screening assessment.
11. Have been treated with any hypoxia-inducible factor-prolyl hydroxylase inhibitor (HIF-PHI) in the 8 weeks prior to randomization
12. have received treatment with an erythropoietic agent, androgenic anabolic steroid, testosterone enanthate or methandrostenolone within 6 weeks prior to screening assessment.
13. a history of significant medical or major surgical procedure within 3 months prior to the screening assessment or elective surgery planned during the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of responding patients | From Baseline to Week 6 or End of Treatment visit
  Responding patient is defined as those with a maximum elevated hemoglobin level greater than 10% of baseline from baseline to five weeks after dosing.

SECONDARY OUTCOMES:
Transfusion treatment rate | From Baseline to Week 6 or End of Treatment visit
  The percentage of subjects who need to receive blood transfusion during the trial
Maximum change in hemoglobin from baseline to 5 weeks post-dose | From Baseline to Week 6 or End of Treatment visit
  Maximum change in hemoglobin from baseline to 5 weeks post-dose
Percentage of visits in which subjects maintained a hemoglobin elevation between >10% and 12.0 g/dL above baseline after reaching 10% of baseline | From Baseline to Week 6 or at End of Treatment visit
  Percentage of visits in which subjects maintained a hemoglobin elevation between >10% and 12.0 g/dL above baseline after reaching 10% of baseline
Percentage of patients who achieve a greater than 10% increase in hemoglobin over baseline during treatment | From Baseline to Week 6 or at End of Treatment visit
  Percentage of patients who achieve a greater than 10% increase in hemoglobin over baseline during treatment
Percentage of subjects requiring blood transfusions during the trial | From Baseline to Week 6 or at End of Treatment visit
  Percentage of subjects requiring blood transfusions during the trial

CONTACTS AND LOCATIONS:
Overall Officials: Yusha Zhu, MD, PhD, Study Director — Kind Pharmaceuticals LLC

IPD SHARING:
Plan to Share IPD: No